CLINICAL TRIAL: NCT06385756
Title: Effect of Amobarbital Sodium Combined With Low-dose Propofol on Hemodynamics During Induction and Perioperative Adverse Reactions in Gynecological Laparoscopic Surgery
Brief Title: Effect of Amobarbital Sodium Combined With Low-dose Propofol on Hemodynamics During Induction and Perioperative Adverse Reactions
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Xuebi Tian, Clinical Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJ-IRB202403020
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Amobarbital Sodium; Hemodynamics Instability
Keywords: Anesthesia induction; Perioperative Adverse Reactions; Gynecological Laparoscopic Surgery
MeSH Terms: interventions — Amobarbital; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- amobarbital-propofol group (Experimental): Participants were given amobarbital sodium 1 mg/kg 1 min before induction and propofol 1.5mg /kg following.
  Interventions: Drug: Amobarbital; Drug: Propofol
- propofol group (Placebo Comparator): The propofol group was given the same volume of normal saline 1 min before induction, followed by propofol 2.5mg /kg.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Amobarbital — Participants with gynecological laparoscopic surgery who met the trial inclusion criteria were randomly divided into 2 groups. After entering the room, peripheral intravenous infusion was opened and oxygen was absorbed by the mask for 5 L/min. Mean arterial pressure, heart rate and oxygen saturation were routinely monitored. After positioning, the amobarbital-propofol group was given amobarbital sodium 1 mg/kg 1 min before induction, followed by Sufentanil 0.5ug /kg, cisatracurium 0.2mg /kg, penehyclidine hydrochloride 0.01mg /kg, propofol 1.5mg /kg for general anesthesia induction. The propofol group was given the same volume of normal saline 1 min before anesthesia induction, followed by Sufentanil 0.5ug /kg, cisatracurium 0.2mg /kg, penehyclidine hydrochloride 0.01mg /kg, propofol 2.5mg /kg.
  Arms: amobarbital-propofol group
Drug: Propofol — propofol

SUMMARY:
At present, there are limited data on perioperative efficacy of barbiturates at home and abroad. The purpose of this clinical trial is to observe the effects of amobarbital sodium combined with low-dose propofol on hemodynamics during induction and perioperative adverse reactions in gynecological laparoscopic surgery patients, and to provide a more reasonable, safe and comfortable anesthesia program for female patients who undergoing laparoscopic surgery.

The main questions it aims to answer are:

* whether the combination of the two results on more stable hemodynamics during induction in gynecological laparoscopic surgery patients;
* whether the incidence of perioperative oxidative stress and inflammation and postoperative nausea and vomiting（ponv） improved after the use of the two combinations of anesthesia induction.

Participants will:

* Induction of anesthesia with the experimental drug or placebo；
* 5 ml of venous blood was retained before, after, and 1 day after surgery for follow-up determination of serum associated factor levels；
* To record their vital signs at any point during the anaesthetic process; Serum serological indexes related to oxidative stress and inflammation were determined. The agitation during the recovery period was recorded. The incidence and severity of ponv were recorded at 2h, 2-6h, and 6-24h postoperatively, and the use of palonosetron was also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 40~60 years old；
* ASA Class I to II；
* The operation time was 1h~2h；
* BMI 18~25；
* Sign informed consent.

Exclusion Criteria:

* Known allergy to narcotic drugs used in this study;
* Severe pulmonary insufficiency;
* Abnormal liver and kidney function；
* History of severe anemia and hematoporphyrin；
* History of asthma;
* Uncontrolled high blood pressure or diabetes;
* Pregnant and lactating women；
* Accompanied by cognitive impairment or inability to communicate.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure (MAP) during Induction of anesthesia | Up to 3 hours
  MAP was recorded as the main index of hemodynamics during anesthesia induction

SECONDARY OUTCOMES:
MAP at different time points | Up to 3 hours
  MAP at different time points (including before induction, tracheal intubation, cutting the skin, extubation)
Incidence of postoperative nausea and vomiting (ponv) | 24 hours
  The incidence of perioperative adverse reactions (ponv) was recorded